CLINICAL TRIAL: NCT00385671
Title: An Open-Label, Randomized Comparison of Duloxetine, Pregabalin, and the Combination of Duloxetine and Gabapentin Among Patients With Inadequate Response to Gabapentin for the Management of Diabetic Peripheral Neuropathic Pain
Brief Title: An Open-Label Comparison of Duloxetine to Other Alternatives for the Management of Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10822; F1J-US-HMEZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride; Pregabalin; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pregabalin (Active Comparator): Pregabalin (PGB) 50 milligram (mg) three times a day (TID) (US & Germany) or 75 mg twice daily (BID) (Canada), orally (PO) for 2 weeks, then PGB 100 mg TID (US & Germany) or 150 mg BID (Canada), PO for 10 weeks.
  Interventions: Drug: pregabalin
- Duloxetine (Experimental): Duloxetine (DLX) 30 milligram (mg) once daily (QD), orally (PO) for 1 week, then DLX 60 mg QD, PO for 11 weeks.
  Interventions: Drug: duloxetine hydrochloride
- Gabapentin + Duloxetine (Experimental): Stable Gabapentin (GAB) + Duloxetine (DLX) 30 milligram (mg) once daily (QD), orally (PO) for 1 week, then stable GAB + DLX 60 mg QD, PO for 11 weeks.
  Interventions: Drug: duloxetine hydrochloride; Drug: gabapentin

INTERVENTIONS:
Drug: duloxetine hydrochloride — Duloxetine (DLX) once daily (QD), orally (PO)
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine; Gabapentin + Duloxetine
Drug: pregabalin — Pregabalin (PGB) orally (PO)
  Arms: Pregabalin
Drug: gabapentin — Stable Gabapentin (GAB) (participants will remain on the same dose of gabapentin at which they entered the study)
  Arms: Gabapentin + Duloxetine

SUMMARY:
To test the non-inferiority of duloxetine monotherapy as a treatment for the management of diabetic peripheral neuropathic pain as compared to pregabalin treatment among patients who have not had an adequate response to gabapentin.

ELIGIBILITY:
Inclusion Criteria:

* You must have been diagnosed with Diabetic Neuropathic Pain
* Patient has an average daily pain score greater than or equal to 4 on an 11-point Likert scale, and patient or provider feel that a change from the current gabapentin therapy for pain management is warranted
* Patient is currently treated with gabapentin greater than or equal to 900 milligram/day, has been prescribed the current dose for at least 4 weeks, and has been at least 80% compliant with dosing, according to patient report
* Patient must agree not to change dose of gabapentin between Visits 1 and 2
* You must have stable glycemic control

Exclusion Criteria:

* Are judged prior to randomization to be at suicidal risk as defined by a score of 2 or greater on question 9 of the Beck Depression Inventory-II (BDI-II)
* Current diagnosis or history of hemangiosarcoma
* Patients with New York Heart Association Class III or IV symptoms of congestive heart failure
* Patients with uncontrolled narrow-angle glaucoma
* Presence of a current seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cromwell, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midvale, Utah
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siegen

REFERENCES:
- [Result] Tanenberg RJ, Irving GA, Risser RC, Ahl J, Robinson MJ, Skljarevski V, Malcolm SK. Duloxetine, pregabalin, and duloxetine plus gabapentin for diabetic peripheral neuropathic pain management in patients with inadequate pain response to gabapentin: an open-label, randomized, noninferiority comparison. Mayo Clin Proc. 2011 Jul;86(7):615-26. doi: 10.4065/mcp.2010.0681. PMID 21719618
- [Derived] Irving G, Tanenberg RJ, Raskin J, Risser RC, Malcolm S. Comparative safety and tolerability of duloxetine vs. pregabalin vs. duloxetine plus gabapentin in patients with diabetic peripheral neuropathic pain. Int J Clin Pract. 2014 Sep;68(9):1130-40. doi: 10.1111/ijcp.12452. Epub 2014 May 18. PMID 24837444
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Started | 134 | 138 | 135
Completed | 96 | 87 | 99
Not Completed | 38 | 51 | 36
Not completed — Adverse Event | 14 | 27 | 18
Not completed — Lack of Efficacy | 5 | 9 | 5
Not completed — Lost to Follow-up | 6 | 6 | 5
Not completed — Physician Decision | 2 | 1 | 2
Not completed — Protocol Violation | 5 | 2 | 1
Not completed — Sponsor Decision | 2 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine | Total
Number analyzed (Participants) | 134 | 138 | 135 | 407
Age Continuous [Mean (Standard Deviation); unit: years] | 61.89 (10.70) | 60.94 (10.18) | 61.85 (10.84) | 61.56 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 52 | 165
  Male | 76 | 83 | 83 | 242
Race/Ethnicity, Customized [Number; unit: participants]
  Native American | 1 | 1 | 1 | 3
  East Asian | 0 | 0 | 2 | 2
  Hispanic | 9 | 15 | 9 | 33
  Black or African American | 13 | 9 | 11 | 33
  White | 111 | 110 | 112 | 333
  West Asian | 0 | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 104 | 112 | 109 | 325
  Germany | 22 | 20 | 21 | 63
  Canada | 5 | 4 | 3 | 12
  Puerto Rico | 3 | 2 | 2 | 7
Duration of Diabetes [Mean (Standard Deviation); unit: months] | 150.26 (131.60) | 147.14 (116.04) | 119.82 (93.38) | 139.09 (115.24)
Duration of Diabetic Peripheral Neuropathic Pain [Mean (Standard Deviation); unit: months] — Duration of Diabetic Peripheral Neuropathic Pain Since Onset.
  months | 51.54 (40.96) | 58.08 (57.57) | 50.32 (41.93) | 53.34 (47.51)
Michigan Neuropathy Screening Instrument (MNSI) Physical Assessment - Total Score [Mean (Standard Deviation); unit: units on a scale] — Assesses degree of neuropathy. Responses to 13 out of 15 items are added to obtain total score. Responses of "yes" to items 1,2,3,5,6,8,9,11,12,14,15 are each counted as one point. A "no" response on items 7 and 13 counts as 1 point. Items 4 and 10 are not included in scoring. Total scores range from 0 (no neuropathy) to 13 (severe neuropathy).
  units on a scale | 5.91 (1.56) | 5.73 (1.58) | 5.94 (1.56) | 5.86 (1.56)
Types of Diabetes Mellitus [Number; unit: participants]
  Type I | 13 | 9 | 9 | 31
  Type II | 121 | 129 | 126 | 376
Weekly mean of 24 hour average pain severity [Mean (Standard Deviation); unit: units on a scale] — This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the average pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries.
  units on a scale | 5.69 (1.43) | 5.81 (1.51) | 5.78 (1.47) | 5.76 (1.47)
Beck Depression Inventory (BDI) Total Score [Mean (Standard Deviation); unit: units on a scale] — A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
  units on a scale | 9.45 (8.53) | 9.10 (7.20) | 10.71 (8.42) | 9.74 (8.07)
Weekly mean of the daily worst pain severity [Mean (Standard Deviation); unit: units on a scale] — This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the daily worst pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries.
  units on a scale | 6.92 (1.56) | 7.12 (1.46) | 7.05 (1.48) | 7.03 (1.50)
Weekly mean of nighttime pain severity [Mean (Standard Deviation); unit: units on a scale] — This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the daily nighttime pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries.
  units on a scale | 5.64 (2.06) | 5.86 (1.74) | 5.55 (2.11) | 5.69 (1.97)
Leeds Sleep Evaluation Questionnaire (LSEQ) [Mean (Standard Deviation); unit: units on a scale] — The LSEQ assesses the effects of psychoactive compounds on sleep and early morning behavior. Participants mark a series of 100 mm line analogue scales, indicating the direction and magnitude of any changes in behavioral state they experience following administration of the drug. Scores are represented in millimeters, higher scores indicate better sleep and better early morning behvior. Subscale score ranges: going to sleep=0-300, quality of sleep=0-200, awakening=0-200, behavior following wakefullness=0-300.
  units on a scale
    Awakening Subscale | 93.95 (41.55) | 88.63 (40.75) | 86.70 (42.46) | 89.75 (41.59)
    Behavior Following Wakefulness Subscale | 132.22 (69.22) | 128.87 (65.53) | 131.55 (69.61) | 130.88 (67.98)
    Getting to Sleep Subscale | 138.62 (59.68) | 137.61 (62.91) | 145.22 (64.73) | 140.45 (62.40)
    Quality of Sleep Subscale | 95.54 (44.08) | 95.89 (46.82) | 97.01 (45.39) | 96.15 (45.34)
Sheehan Disability Scale (SDS) Global Functional Impairment Total Score [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life.
  units on a scale | 11.44 (8.72) | 13.49 (9.00) | 12.69 (7.92) | 12.55 (8.58)
Clayton Sexual Functioning Questionnaire (CSFQ) [Mean (Standard Deviation); unit: units on a scale] — The CSFQ is a 14-item subject-rated scale designed to assess changes in sexual activity and functioning. The CSFQ is a structured interview/questionnaire, which is designed to measure medication related changes in sexual functioning. The CSFQ measures five dimensions of sexual behavior: pleasure; desire/frequency; desire/interest; arousal; and orgasm. The CSFQ total score is also obtained across all 5 dimensions and ranges from 14 to 70. Subscale score ranges: desire/frequency=2-10; desire/interest=3-15; pleasure=1-5; arousal=3-15; orgasm=3-15. Higher scores indicate greater changes.
  units on a scale
    male participants - total | 40.41 (9.01) | 38.81 (9.50) | 39.25 (9.75) | 39.46 (9.42)
    female participants - total | 35.21 (11.68) | 36.69 (10.43) | 34.45 (10.09) | 35.43 (10.73)
    male participants - arousal | 7.19 (3.08) | 6.35 (2.88) | 6.41 (3.12) | 6.64 (3.04)
    female participants - arousal | 6.64 (3.20) | 7.00 (2.72) | 6.47 (3.09) | 6.70 (3.01)
    male participants - desire/frequency | 5.32 (1.73) | 5.09 (1.77) | 5.15 (1.96) | 5.18 (1.82)
    female participants - desire/frequency | 3.79 (1.85) | 4.27 (1.83) | 3.74 (1.59) | 3.93 (1.77)
    male participants - desire/interest | 7.71 (2.56) | 7.91 (2.72) | 8.06 (2.84) | 7.90 (2.71)
    female participants - desire/interest | 5.96 (3.01) | 5.97 (2.42) | 5.72 (2.43) | 5.89 (2.63)
    male participants - orgasm | 7.77 (2.93) | 7.21 (2.85) | 7.51 (3.06) | 7.49 (2.94)
    female participants - orgasm | 6.98 (3.75) | 8.23 (3.94) | 7.53 (3.83) | 7.56 (3.84)
    male participants - pleasure | 2.43 (1.23) | 2.50 (1.22) | 2.30 (1.11) | 2.41 (1.19)
    female participants - pleasure | 2.06 (1.19) | 2.23 (1.18) | 2.06 (1.13) | 2.12 (1.16)
Comorbidity with Generalized Anxiety Disorder (GAD) [Number; unit: participants] — Frequency of current comorbid Generalized Anxiety Disorder-Text-Revised (DSM-IV-TR) based on specific modules of the Mini-International Neuropsychiatric Interview (MINI), a short, structured diagnostic interview developed for DSM-IV psychiatric disorders.
  participants
    Yes | 3 | 0 | 1 | 4
    No | 131 | 138 | 134 | 403
Comorbidity with Major Depressive Disorder (MDD) [Number; unit: participants] — Frequency of current comorbid Major Depressive Disorder-Text revision (DSM-IV-TR) based on specific modules of the Mini-International Neuropsychiatric Interview (MINI), a short, structured diagnostic interview developed for DSM-IV psychiatric disorders.
  participants
    Yes | 4 | 3 | 4 | 11
    No | 130 | 135 | 131 | 396

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 12 Weeks in Weekly Mean of Daily 24 Hour Average Pain Score, Pregabalin Compared With Duloxetine
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the average pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: All randomized participants with a baseline value and at least 1 non-missing post-baseline value (modified intent-to-treat population) were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine
Number analyzed (Participants) | 93 | 77
units on a scale | -2.12 (0.19) | -2.62 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Null hypothesis: no difference in mean change from baseline to 12 weeks in weekly mean of daily 24 hour average pain score between pregabalin & duloxetine treatments. Sample size: 125 participants/treatment, 6% increase for 400 planned enrollees. 92% power with 1-sided 97.5% confidence interval; mean change in duloxetine group, -2.7; in pregabalin group, -2.5; standard deviation, 2.3; margin of non-inferiority: -0.8; Test type: Non-Inferiority or Equivalence — Basis of non-inferiority margin (maximum disadvantage for duloxetine compared to pregabalin not considered meaningful): In 3 previous placebo-controlled trials of duloxetine in DPNP, in the subgroup of patients that had been treated with gabapentin prior to entry, the estimated mean change in pain at Week 12 was -2.74 for duloxetine and -1.09 for placebo, an advantage of about 1.65. The non-inferiority margin represents about half of this previous treatment effect in a similar population; p = 0.076, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons and 0.10 for tests of interaction; Change=Treatment+InvestigatorGroup+Week+Baseline+Treatment*Week+Baseline*Week, Kenward-Roger approximation was used; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.05 to 1.04]

2. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Weekly Mean of Daily 24 Hour Average Pain Score, Duloxetine Compared With Duloxetine+Gabapentin
Description: as for outcome 1
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Gabapentin + Duloxetine | Duloxetine
Number analyzed (Participants) | 86 | 77
units on a scale | -2.39 (0.20) | -2.62 (0.21)
Statistical Analysis 1: Comparison: Gabapentin + Duloxetine vs Duloxetine; Null hypothesis: no difference in mean change from baseline to 12 weeks in weekly mean of daily 24 hour average pain score between duloxetine & duloxetine+gabapentin treatments. Sample size: 125 participants/treatment, 6% increase for 400 planned enrollees. 92% power with 1-sided 97.5% confidence interval; mean change in duloxetine group, -2.7; in pregabalin group, -2.5; standard deviation, 2.3; margin of non-inferiority: -0.8; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.417, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Change=Treatment+InvestigatorGroup+Week+Baseline+Treatment*Week+Baseline*Week, Kenward-Roger approximation was used; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.32 to 0.78]

3. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Weekly Mean of Nighttime Pain Severity
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the daily nighttime pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
units on a scale | -2.30 (0.21) | -2.71 (0.22) | -2.49 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in Weekly mean of nighttime pain severity; Test type: Superiority or Other; p = 0.463, Mixed Models Analysis — P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; Change=Treatment+InvestigatorGroup+Week+Baseline+Treatment*Week+Baseline*Week; denominator degrees of freedom, Kenward-Rogers approximation
Statistical Analysis 2: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Weekly mean of nighttime pain severity; Test type: Superiority or Other; p = 0.520, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Weekly mean of nighttime pain severity; Test type: Superiority or Other; p = 0.463, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Weekly Mean of the Daily Worst Pain Severity Score
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the daily worst pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
units on a scale | -2.59 (0.22) | -3.08 (0.24) | -2.86 (0.23)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in weekly mean of the daily worst pain severity score; Test type: Superiority or Other; p = 0.389, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in weekly mean of the daily worst pain severity score; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in weekly mean of the daily worst pain severity score; Test type: Superiority or Other; p = 0.489, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Clinical Global Impression of Severity Scale (CGI Severity)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 117 | 125 | 120
units on a scale
  baseline | 4.27 (0.85) | 4.47 (0.90) | 4.40 (0.79)
  change | -1.06 (0.10) | -1.16 (0.10) | -1.13 (0.10)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in CGI severity; Test type: Superiority or Other; p = 0.602, t-test, 2 sided — P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; Analysis of Covariance model and t-tests: Change=InvestigatorGroup+Baseline+Treatment. Last-observation-carried-forward imputation was used; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.20 to 0.35]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in CGI severity; Test type: Superiority or Other; p = 0.469, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.17 to 0.37]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in CGI severity; Test type: Superiority or Other; p = 0.841, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.24 to 0.30]

6. Secondary Outcome: Patient's Global Impression of Improvement Scale (PGI - Improvement) at 12 Weeks
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 122 | 125 | 121
units on a scale | 3.03 (1.19) | 3.01 (1.68) | 2.83 (1.27)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in PGI-Improvement at 12 weeks; Test type: Superiority or Other; p = 0.276, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; Analysis of Variance model and t-tests: Endpoint = InvestigatorGroup + Treatment. Last-observation-carried-forward imputation was implemented; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.16 to 0.55]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in PGI-Improvement at 12 weeks; Test type: Superiority or Other; p = 0.929, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.33 to 0.37]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in PGI-Improvement at 12 weeks; Test type: Superiority or Other; p = 0.313, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.53 to 0.17]

7. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Severity: 24-hour Average Pain
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 5.53 (1.87) | 5.65 (1.72) | 5.75 (1.76)
  change | -1.80 (0.20) | -2.44 (0.21) | -2.29 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-Severity: 24-hour average pain; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.06 to 1.04]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-Severity: 24-hour average pain; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [0.08 to 1.20]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-Severity: 24-hour average pain; Test type: Superiority or Other; p = 0.602, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.41 to 0.70]

8. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Severity: Worst Pain
Description: A self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 6.73 (2.01) | 6.87 (2.06) | 7.00 (1.83)
  change | -2.34 (0.23) | -3.02 (0.25) | -2.64 (0.23)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-severity: worst pain; Test type: Superiority or Other; p = 0.353, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.34 to 0.94]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-severity: worst pain; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.03 to 1.34]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-Severity: Worst Pain; Test type: Superiority or Other; p = 0.244, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.27 to 1.04]

9. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Severity: Least Pain
Description: A self-reported scale that measures the severity of pain based on the least pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 4.23 (2.28) | 4.18 (2.11) | 4.07 (2.14)
  change | -1.27 (0.19) | -1.55 (0.20) | -1.54 (0.19)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-Severity: Least Pain; Test type: Superiority or Other; p = 0.298, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.25 to 0.80]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-Severity: Least Pain; Test type: Superiority or Other; p = 0.304, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.25 to 0.81]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-severity: least pain; Test type: Superiority or Other; p = 0.989, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.53 to 0.54]

10. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Severity: Pain Right Now
Description: A self-reported scale that measures the severity of pain based on the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 4.98 (2.33) | 5.03 (2.30) | 5.36 (2.18)
  change | -1.77 (0.21) | -2.24 (0.22) | -2.19 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-severity: pain right now; Test type: Superiority or Other; p = 0.145, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.14 to 0.97]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.112, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.11 to 1.03]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.865, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.52 to 0.62]

11. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference: With General Activity
Description: A self-reported scale that measures the interference of pain in the past 24 hours on general activity. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 4.24 (2.67) | 5.03 (2.65) | 5.03 (2.48)
  change | -1.51 (0.22) | -2.38 (0.23) | -1.86 (0.22)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with general activity; Test type: Superiority or Other; p = 0.263, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.26 to 0.95]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with general activity; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [0.24 to 1.49]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with general activity; Test type: Superiority or Other; p = 0.102, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.10 to 1.13]

12. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference With Mood
Description: A self-reported scale that measures the interference of pain in the past 24 hours on mood. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 3.42 (2.73) | 4.08 (2.66) | 4.10 (2.67)
  change | -1.46 (0.21) | -1.85 (0.23) | -1.43 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with mood; Test type: Superiority or Other; p = 0.922, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.61 to 0.55]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with mood; Test type: Superiority or Other; p = 0.195, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.20 to 0.99]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with mood; Test type: Superiority or Other; p = 0.162, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.17 to 1.02]

13. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference With Walking Ability
Description: A self-reported scale that measures the interference of pain in the past 24 hours on walking ability. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 5.25 (2.72) | 5.52 (2.85) | 5.79 (2.53)
  change | -1.88 (0.24) | -2.56 (0.26) | -2.09 (0.24)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with walking ability; Test type: Superiority or Other; p = 0.541, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.46 to 0.87]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with walking ability; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-0.00 to 1.36]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with walking ability; Test type: Superiority or Other; p = 0.173, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.21 to 1.15]

14. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference With Normal Work
Description: A self-reported scale that measures the interference of pain in the past 24 hours on normal work. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 130 | 126
units on a scale
  baseline | 4.61 (2.86) | 4.98 (2.86) | 5.15 (2.54)
  change | -1.63 (0.24) | -1.86 (0.25) | -1.88 (0.24)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Weekly BPI-interference with normal work; Test type: Superiority or Other; p = 0.451, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.40 to 0.90]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with normal work; Test type: Superiority or Other; p = 0.485, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.43 to 0.90]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with normal work; Test type: Superiority or Other; p = 0.969, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.68 to 0.65]

15. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference With Relations With Other People
Description: A self-reported scale that measures the interference of pain in the past 24 hours on relations with other people. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 2.96 (2.68) | 3.08 (2.72) | 3.29 (2.58)
  change | -0.97 (0.21) | -1.27 (0.22) | -1.17 (0.21)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Weekly BPI-interference with relations with other people; Test type: Superiority or Other; p = 0.479, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.36 to 0.76]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with relations with other people; Test type: Superiority or Other; p = 0.301, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.27 to 0.87]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with relations with other people; Test type: Superiority or Other; p = 0.731, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.47 to 0.67]

16. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference With Sleep
Description: A self-reported scale that measures the interference of pain in the past 24 hours on sleep. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 4.91 (2.87) | 4.97 (2.94) | 5.40 (2.81)
  change | -2.29 (0.24) | -2.12 (0.26) | -2.50 (0.24)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with sleep; Test type: Superiority or Other; p = 0.528, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.45 to 0.87]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with sleep; Test type: Superiority or Other; p = 0.626, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.84 to 0.51]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with sleep; Test type: Superiority or Other; p = 0.270, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.06 to 0.30]

17. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Interference With Enjoyment of Life
Description: A self-reported scale that measures the interference of pain in the past 24 hours on enjoyment of life. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 4.38 (3.08) | 4.63 (2.96) | 5.02 (2.68)
  change | -1.82 (0.22) | -2.09 (0.24) | -2.33 (0.23)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with enjoyment of life; Test type: Superiority or Other; p = 0.098, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.10 to 1.13]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI-interference with enjoyment of life; Test type: Superiority or Other; p = 0.383, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.35 to 0.90]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI-interference with enjoyment of life; Test type: Superiority or Other; p = 0.452, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.86 to 0.39]

18. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Brief Pain Inventory (BPI) - Mean Interference Score
Description: The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 128 | 130 | 126
units on a scale
  baseline | 4.25 (2.34) | 4.61 (2.36) | 4.83 (2.13)
  change | -1.62 (0.20) | -2.00 (0.21) | -1.90 (0.20)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI mean interference score; Test type: Superiority or Other; p = 0.309, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.26 to 0.82]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BPI mean interference score; Test type: Superiority or Other; p = 0.174, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.17 to 0.93]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BPI mean interference score; Test type: Superiority or Other; p = 0.717, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.45 to 0.65]

19. Secondary Outcome: Number of Participants With ≥ 30% Reduction in the Weekly Mean 24 Hour Average Pain Score at 12 Weeks
Description: This is a nominal outcome reflecting whether or not a clinically-important efficacy outcome was achieved at endpoint. It is based on a comparison between baseline and endpoint scores on an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Used were the weekly mean of the scores of the average pain severity over the last 24 hours. The weekly averages were based on daily assessments recorded by patients in their diaries.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
participants | 65 | 68 | 72
Statistical Analysis 1: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with ≥ 30% reduction in the weekly mean 24 hour average pain score at 12 weeks; Test type: Superiority or Other; p = 0.975, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; Treatments were compared with stratification defined by InvestigatorGroup. Last-observation-carried-forward imputation was implemented
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with ≥ 30% reduction in the weekly mean 24 hour average pain score at 12 weeks; Test type: Superiority or Other; p = 0.448, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with ≥ 30% reduction in the weekly mean 24 hour average pain score at 12 weeks; Test type: Superiority or Other; p = 0.280, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]

20. Secondary Outcome: Number of Patients With a Reduction of ≥ 50% in Weekly Mean of 24 Hour Average Pain Score
Description: as for outcome 19
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
participants | 48 | 50 | 47
Statistical Analysis 1: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of patients with a reduction of ≥ 50% in Weekly mean of 24 hour average pain score; Test type: Superiority or Other; p = 0.548, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of patients with a reduction of ≥ 50% in Weekly mean of 24 hour average pain score; Test type: Superiority or Other; p = 0.599, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference in the number of patients with a reduction of ≥ 50% in Weekly mean of 24 hour average pain score; Test type: Superiority or Other; p = 1.00, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]

21. Secondary Outcome: Number of Participants With a ≥ 2-points Reduction on the Weekly Average of the Daily 24-hour Average Pain Scale at 12 Weeks
Description: as for outcome 19
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
participants | 59 | 64 | 68
Statistical Analysis 1: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of Participants with a ≥ 2-points reduction on the weekly average of the daily 24-hour average pain scale at 12 Weeks; Test type: Superiority or Other; p = 0.905, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of Participants with a ≥ 2-points reduction on the weekly average of the daily 24-hour average pain scale at 12 Weeks; Test type: Superiority or Other; p = 0.368, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin + Duloxetine; [analysis description as in outcome 21, analysis 2]; Test type: Superiority or Other; p = 0.200, Mantel Haenszel — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 19, analysis 1]

22. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Leeds Sleep Evaluation Questionnaire (LSEQ) Subscales of Ease of Going to Sleep (GTS), Awakening (AFS), and Behavior Following Wakefulness (BFW), Quality of Sleep (QOS)
Description: The LSEQ assesses the effects of psychoactive compounds on sleep and early morning behavior. Participants mark a series of 100 mm line analogue scales, indicating the direction and magnitude of any changes in behavioral state they experience following administration of the drug. Scores are represented in millimeters, higher scores indicate better sleep and better early morning behavior. Subscale score ranges: GTS=0-300, QOS=0-200, AFS=0-200, BFW=0-300. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 124 | 119 | 118
units on a scale
  GTS, n=122, n=119, n=118 | 10.96 (4.83) | 17.40 (5.06) | 14.75 (4.92)
  QOS, n=121, n=118, n=118 | 9.32 (4.01) | 7.39 (4.24) | 9.64 (4.06)
  AFS, n=122, n=118, n=118 | 10.02 (3.71) | 8.14 (3.92) | 11.86 (3.73)
  BFW, n=124, n=115, n=118 | 19.67 (5.65) | 21.04 (6.03) | 14.33 (5.77)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ GTS scores; Test type: Superiority or Other; p = 0.572, Mixed Models Analysis — P-value is for GTS. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 weeks in LSEQ GTS scores; Test type: Superiority or Other; p = 0.345, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ GTS scores; Test type: Superiority or Other; p = 0.699, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ QOS scores; Test type: Superiority or Other; p = 0.954, Mixed Models Analysis — P-value is for QOS. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in LSEQ QOS scores; Test type: Superiority or Other; p = 0.734, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 4]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ QOS; Test type: Superiority or Other; p = 0.693, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 4]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ AFS scores; Test type: Superiority or Other; p = 0.720, Mixed Models Analysis — P-value is for AFS. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in LSEQ AFS scores; Test type: Superiority or Other; p = 0.722, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 7]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ AFS scores; Test type: Superiority or Other; p = 0.480, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 7]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ BFW scores; Test type: Superiority or Other; p = 0.498, Mixed Models Analysis — P-value is for BFW. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in LSEQ BFW scores; Test type: Superiority or Other; p = 0.865, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 10]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in LSEQ BFW scores; Test type: Superiority or Other; p = 0.408, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 10]; [statistical method as in outcome 3, analysis 1]

23. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Sheehan Disability Scale (SDS) - Total Score and Scores for Items 1 to 3
Description: The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total scores range from 0 to 30, higher values indicate greater disruption in the patient's life. Item 1 assesses the effect of the patient's symptoms on their work/school schedule, Item 2 on their social life/leisure activities, and Item 3 on their family life/home responsibilities. Subscales scores range: 0-10, higher values indicate greater disruption in the patient's life. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 118 | 124 | 119
units on a scale
  Total | -4.96 (0.66) | -3.47 (0.65) | -4.54 (0.66)
  Item 1 | -1.96 (0.31) | -1.21 (0.33) | -1.95 (0.32)
  Item 2 | -1.64 (0.24) | -1.12 (0.23) | -1.53 (0.24)
  Item 3 | -1.70 (0.22) | -1.17 (0.22) | -1.54 (0.22)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS total score; Test type: Superiority or Other; p = 0.635, t-test, 2 sided — P-value is for total. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-2.18 to 1.33]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in SDS total score; Test type: Superiority or Other; p = 0.092, t-test, 2 sided — [p-value comment as in outcome 23, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-3.24 to 0.24]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS total score; Test type: Superiority or Other; p = 0.221, t-test, 2 sided — [p-value comment as in outcome 23, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-2.80 to 0.65]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS Item 1 score; Test type: Superiority or Other; p = 0.974, t-test, 2 sided — P-value is for item 1. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.88 to 0.85]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in SDS Item 1 score; Test type: Superiority or Other; p = 0.093, t-test, 2 sided — [p-value comment as in outcome 23, analysis 4]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.63 to 0.13]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS Item 1 score; Test type: Superiority or Other; p = 0.091, t-test, 2 sided — [p-value comment as in outcome 23, analysis 4]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.59 to 0.12]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS Item 2 score; Test type: Superiority or Other; p = 0.733, t-test, 2 sided — P-value is for item 2. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.75 to 0.52]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in SDS item 2 score; Test type: Superiority or Other; p = 0.102, t-test, 2 sided — [p-value comment as in outcome 23, analysis 7]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.15 to 0.11]
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS item 2 score; Test type: Superiority or Other; p = 0.193, t-test, 2 sided — [p-value comment as in outcome 23, analysis 7]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-1.04 to 0.21]
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS item 3 score; Test type: Superiority or Other; p = 0.584, t-test, 2 sided — P-value is for item 3. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.76 to 0.43]
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in SDS item 3 score; Test type: Superiority or Other; p = 0.077, t-test, 2 sided — [p-value comment as in outcome 23, analysis 10]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.12 to 0.06]
Statistical Analysis 12: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in SDS item 3 score; Test type: Superiority or Other; p = 0.221, t-test, 2 sided — [p-value comment as in outcome 23, analysis 10]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.95 to 0.22]

24. Secondary Outcome: Summary of Adverse Events and Serious Adverse Events Leading to Discontinuation
Time Frame: baseline through 12 weeks
Population: All participants who were enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 134 | 138 | 135
participants
  Nausea | 0 | 4 | 4
  Peripheral Oedema | 5 | 0 | 0
  Insomnia | 0 | 4 | 0
  Somnolence | 1 | 2 | 0
  Anxiety | 0 | 1 | 1
  Dizziness | 0 | 0 | 2
  Dysuria | 0 | 2 | 0
  Headache | 0 | 2 | 0
  Hyperhidrosis | 0 | 1 | 1
  Sedation | 1 | 0 | 1
  Allergic Oedema | 1 | 0 | 0
  Anorgasmia | 0 | 1 | 0
  Increased Blood Creatine | 0 | 0 | 1
  Increased Blood Glucose | 1 | 0 | 0
  Bruxism | 0 | 1 | 0
  Cerebrovascular Accident | 0 | 1 | 0
  Chest Discomfort | 0 | 0 | 1
  Depression | 0 | 1 | 0
  Dermatitis | 0 | 1 | 0
  Diarrhoea | 0 | 0 | 1
  Dry mouth | 0 | 1 | 0
  Enterovirus Infection | 0 | 0 | 1
  Fatigue | 0 | 1 | 0
  Generalized Oedema | 1 | 0 | 0
  Facial Hypoaesthesia | 1 | 0 | 0
  Lacunar Infarction | 1 | 0 | 0
  Loss of Consciousness | 0 | 1 | 0
  Lymphoma | 0 | 0 | 1
  Mental Impairment | 1 | 0 | 0
  Muscular Weakness | 0 | 0 | 1
  Myoclonus | 0 | 1 | 0
  Pollakiuria | 0 | 0 | 1
  Pulomnary Embolism | 0 | 0 | 1
  Rash | 0 | 0 | 1
  Sleep Disorder | 0 | 1 | 0
  Urticaria | 1 | 0 | 0
  Vomiting | 0 | 1 | 0

25. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) Total Score and Subscale Scores
Description: 14-item subject-rated scale assessing medication related changes in sexual activity + functioning. Structured interview/questionnaire. It measures five dimensions of sexual behavior: pleasure; desire/frequency; desire/interest; arousal; and orgasm. The total score is obtained across all 5 dimensions, ranging from 14 to 70. Subscale score ranges: desire/frequency=2-10; desire/interest=3-15; pleasure=1-5; arousal=3-15; orgasm=3-15. Higher scores = better sexual functioning. Least-squares means: adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 101 | 109 | 109
units on a scale
  male, total; n=62, n=67, n=66 | -0.53 (0.80) | 0.48 (0.77) | 1.29 (0.79)
  female, total; n=39; n=42, n=43 | -0.01 (1.10) | 1.12 (1.10) | -0.61 (1.08)
  male, pleasure; n=64, n=67, n=69 | 0.08 (0.12) | -0.06 (0.11) | 0.13 (0.11)
  female, pleasure; n=40, n=42, n=43 | 0.15 (0.16) | 0.47 (0.16) | -0.09 (0.16)
  male, desire/frequency; n=65, n=67, n=69 | -0.02 (0.16) | 0.06 (0.16) | 0.16 (0.16)
  female, desire/frequency; n=42, n=42, n=43 | 0.21 (0.21) | 0.26 (0.22) | 0.30 (0.21)
  male, desire/interest; n=65, n=67, n=70 | -0.27 (0.24) | -0.19 (0.24) | 0.05 (0.24)
  female, desire/interest; n=42, n=42, n=45 | -0.17 (0.32) | 0.34 (0.33) | 0.01 (0.32)
  male, arousal; n=65, n=67, n=70 | 0.17 (0.26) | 0.52 (0.26) | 0.52 (0.26)
  female, arousal; n=40, n=42, n=45 | -0.11 (0.34) | 0.07 (0.35) | -0.30 (0.33)
  male, orgasm; n=64, n=67, n=69 | -0.39 (0.27) | 0.18 (0.26) | 0.17 (0.26)
  female, orgasm; n=40, n=42, n=43 | 0.31 (0.39) | -0.05 (0.40) | -0.85 (0.39)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) total score; Test type: Superiority or Other; p = 0.096, t-test, 2 sided — P-value is for male, total. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-3.96 to 0.32]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) total score; Test type: Superiority or Other; p = 0.353, t-test, 2 sided — [p-value comment as in outcome 25, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-3.16 to 1.13]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) total score; Test type: Superiority or Other; p = 0.444, t-test, 2 sided — [p-value comment as in outcome 25, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-1.27 to 2.88]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) total score; Test type: Superiority or Other; p = 0.682, t-test, 2 sided — P-value is for female, total. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-2.29 to 3.48]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) total score; Test type: Superiority or Other; p = 0.450, t-test, 2 sided — [p-value comment as in outcome 25, analysis 4]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-4.08 to 1.82]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) total score; Test type: Superiority or Other; p = 0.218, t-test, 2 sided — [p-value comment as in outcome 25, analysis 4]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-4.49 to 1.04]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) pleasure subscore; Test type: Superiority or Other; p = 0.747, t-test, 2 sided — P-value is for male, pleasure. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.36 to 0.26]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) pleasure subscore; Test type: Superiority or Other; p = 0.390, t-test, 2 sided — [p-value comment as in outcome 25, analysis 7]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.18 to 0.45]
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) pleasure subscore; Test type: Superiority or Other; p = 0.228, t-test, 2 sided — [p-value comment as in outcome 25, analysis 7]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.12 to 0.49]
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) pleasure subscore; Test type: Superiority or Other; p = 0.260, t-test, 2 sided — P-value is for female, pleasure. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.18 to 0.67]
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) pleasure subscore; Test type: Superiority or Other; p = 0.141, t-test, 2 sided — [p-value comment as in outcome 25, analysis 10]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.76 to 0.11]
Statistical Analysis 12: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) pleasure subscore; Test type: Superiority or Other; p = 0.007, t-test, 2 sided — [p-value comment as in outcome 25, analysis 10]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.98 to -0.16]
Statistical Analysis 13: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/frequency subscore; Test type: Superiority or Other; p = 0.409, t-test, 2 sided — P-value is for male, desire/frequency. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.61 to 0.25]
Statistical Analysis 14: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/frequency subscore; Test type: Superiority or Other; p = 0.715, t-test, 2 sided — [p-value comment as in outcome 25, analysis 13]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.51 to 0.35]
Statistical Analysis 15: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/frequency subscore; Test type: Superiority or Other; p = 0.641, t-test, 2 sided — [p-value comment as in outcome 25, analysis 13]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.32 to 0.52]
Statistical Analysis 16: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/frequency subscore; Test type: Superiority or Other; p = 0.767, t-test, 2 sided — P-value is for female, desire/frequency. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.64 to 0.47]
Statistical Analysis 17: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/frequency subscore; Test type: Superiority or Other; p = 0.881, t-test, 2 sided — [p-value comment as in outcome 25, analysis 16]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.61 to 0.52]
Statistical Analysis 18: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/frequency subscore; Test type: Superiority or Other; p = 0.885, t-test, 2 sided — [p-value comment as in outcome 25, analysis 16]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.51 to 0.59]
Statistical Analysis 19: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/interest subscore; Test type: Superiority or Other; p = 0.325, t-test, 2 sided — P-value is for male, desire/interest. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.96 to 0.32]
Statistical Analysis 20: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/interest subscore; Test type: Superiority or Other; p = 0.798, t-test, 2 sided — [p-value comment as in outcome 25, analysis 19]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.73 to 0.56]
Statistical Analysis 21: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/interest subscore; Test type: Superiority or Other; p = 0.461, t-test, 2 sided — [p-value comment as in outcome 25, analysis 19]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.39 to 0.87]
Statistical Analysis 22: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/interest subscore; Test type: Superiority or Other; p = 0.670, t-test, 2 sided — p-value is for female, desire/interest. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-1.02 to 0.66]
Statistical Analysis 23: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) desire/interest subscore; Test type: Superiority or Other; p = 0.243, t-test, 2 sided — [p-value comment as in outcome 25, analysis 22]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.37 to 0.35]
Statistical Analysis 24: Comparison: Duloxetine vs Gabapentin + Duloxetine; [analysis description as in outcome 25, analysis 19]; Test type: Superiority or Other; p = 0.423, t-test, 2 sided — [p-value comment as in outcome 25, analysis 22]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.14 to 0.48]
Statistical Analysis 25: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) arousal subscore; Test type: Superiority or Other; p = 0.333, t-test, 2 sided — P-value is for male, arousal. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.04 to 0.35]
Statistical Analysis 26: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) arousal subscore; Test type: Superiority or Other; p = 0.334, t-test, 2 sided — [p-value comment as in outcome 25, analysis 25]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.05 to 0.36]
Statistical Analysis 27: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) arousal subscore; Test type: Superiority or Other; p = 0.990, t-test, 2 sided — [p-value comment as in outcome 25, analysis 25]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.69 to 0.68]
Statistical Analysis 28: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) arousal subscore; Test type: Superiority or Other; p = 0.665, t-test, 2 sided — P-value is for female, arousal. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.70 to 1.09]
Statistical Analysis 29: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) arousal subscore; Test type: Superiority or Other; p = 0.700, t-test, 2 sided — [p-value comment as in outcome 25, analysis 28]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-1.10 to 0.74]
Statistical Analysis 30: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) arousal subscore; Test type: Superiority or Other; p = 0.386, t-test, 2 sided — [p-value comment as in outcome 25, analysis 28]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.23 to 0.48]
Statistical Analysis 31: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) orgasm subscore; Test type: Superiority or Other; p = 0.120, t-test, 2 sided — P-value is for male, orgasm. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.27 to 0.15]
Statistical Analysis 32: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) orgasm subscore; Test type: Superiority or Other; p = 0.119, t-test, 2 sided — [p-value comment as in outcome 25, analysis 31]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.29 to 0.15]
Statistical Analysis 33: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in male participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) orgasm subscore; Test type: Superiority or Other; p = 0.976, t-test, 2 sided — [p-value comment as in outcome 25, analysis 25]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.71 to 0.69]
Statistical Analysis 34: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) orgasm subscore; Test type: Superiority or Other; p = 0.026, t-test, 2 sided — P-value is for female, orgasm. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [0.14 to 2.20]
Statistical Analysis 35: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) orgasm subscore; Test type: Superiority or Other; p = 0.497, t-test, 2 sided — [p-value comment as in outcome 25, analysis 34]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-0.69 to 1.42]
Statistical Analysis 36: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in female participants in mean change from baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) orgasm subscore; Test type: Superiority or Other; p = 0.112, t-test, 2 sided — [p-value comment as in outcome 25, analysis 34]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.80 to 0.19]

26. Secondary Outcome: Categorical Change From Baseline to 12 Weeks in Sexual Functioning Questionnaire (CSFQ) Total Score and Subscale Scores
Description: 14-item subject-rated scale assessing changes in sexual activity and functioning; structured interview/questionnaire, designed to measure medication related changes in sexual functioning. 5 dimensions of sexual behavior: pleasure; desire/frequency; desire/interest; arousal; orgasm. Total score: obtained across all 5 dimensions, ranges from 14 to 70. Subscale scores: desire/frequency=2-10; desire/interest=3-15; pleasure=1-5; arousal=3-15; orgasm=3-15. Higher scores = better sexual functioning. Categories: better=positive change in score; same=no change in score; worse=negative change in score.
Time Frame: baseline, 12 weeks
Population: All randomized participants with a baseline value and at least 1 non-missing post-baseline value (modified intent-to-treat population) and with baseline values within the normal range were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 134 | 138 | 135
participants
  male, total, better; n=62, n=67, n=66 | 24 | 26 | 31
  male, total, same; n=62, n=67, n=66 | 9 | 9 | 11
  male, total, worse; n=62, n=67, n=66 | 29 | 32 | 24
  female, total, better; n=39, n=42, n=43 | 13 | 23 | 18
  female, total, same; n=39, n=42, n=43 | 5 | 5 | 7
  female, total, worse; n=39, n=42, n=43 | 21 | 14 | 18
  male, pleasure, better; n=64, n=67, n=69 | 13 | 11 | 21
  male, pleasure, same; n=64, n=67, n=69 | 39 | 40 | 32
  male, pleasure, worse; n=64, n=67, n=69 | 12 | 16 | 16
  female, pleasure, better; n=40, n=42, n=43 | 10 | 16 | 6
  female, pleasure, same; n=40, n=42, n=43 | 23 | 21 | 32
  female, pleasure, worse; n=40, n=42, n=43 | 7 | 5 | 5
  male, desire/frequency, better; n=65, n=67, n=69 | 12 | 20 | 24
  male, desire/frequency, same; n=65, n=67, n=69 | 36 | 29 | 23
  male, desire/frequency, worse; n=65, n=67, n=69 | 17 | 18 | 22
  female, desire/frequency, better; n=42, n=42, n=43 | 11 | 12 | 12
  female, desire/frequency, same; n=42, n=42, n=43 | 21 | 21 | 24
  female, desire/frequency, worse; n=42, n=42, n=43 | 10 | 9 | 7
  male, desire/interest, better; n=65, n=67, n=70 | 20 | 18 | 26
  male, desire/interest, same; n=65, n=67, n=70 | 19 | 19 | 17
  male, desire/interest, worse; n=65, n=67, n=70 | 26 | 30 | 27
  female, desire/interest, better; n=42, n=42, n=45 | 13 | 18 | 16
  female, desire/interest, same; n=42, n=42, n=45 | 12 | 14 | 17
  female, desire/interest, worse; n=42, n=42, n=45 | 17 | 10 | 12
  male, arousal, better; n=65, n=67, n=70 | 20 | 24 | 23
  male, arousal, same; n=65, n=67, n=70 | 28 | 29 | 33
  male, arousal, worse; n=65, n=67, n=70 | 17 | 14 | 14
  female, arousal, better; n=40, n=42, n=45 | 11 | 18 | 15
  female, arousal, same; n=40, n=42, n=45 | 14 | 10 | 16
  female, arousal, worse; n=40, n=42, n=45 | 15 | 14 | 14
  male, orgasm, better; n=64, n=67, n=69 | 12 | 18 | 17
  male, orgasm, same; n=64, n=67, n=69 | 29 | 31 | 29
  male, orgasm, worse; n=64, n=67, n=69 | 23 | 18 | 23
  female, orgasm, better; n=40, n=42, n=43 | 15 | 17 | 11
  female, orgasm, same; n=40, n=42, n=43 | 13 | 13 | 16
  female, orgasm, worse; n=40, n=42, n=43 | 12 | 12 | 16
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of male participants with a categorical change in total score from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.486, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of male participants with a categorical change in total score from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.983, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of male participants with a categorical change in total score from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.411, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of female participants with a categorical change in total score from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.554, Chi-squared — [p-value comment as in outcome 25, analysis 4]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of female participants with a categorical change in total score from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.128, Chi-squared — [p-value comment as in outcome 25, analysis 4]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of female participants with a categorical change in total score from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.488, Chi-squared — [p-value comment as in outcome 25, analysis 4]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of male participants with a categorical change in pleasure subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.226, Chi-squared — [p-value comment as in outcome 25, analysis 7]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of male participants with a categorical change in pleasure subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.710, Chi-squared — [p-value comment as in outcome 25, analysis 7]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of male participants with a categorical change in pleasure subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.133, Chi-squared — [p-value comment as in outcome 25, analysis 7]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of female participants with a categorical change in pleasure subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.257, Chi-squared — [p-value comment as in outcome 25, analysis 10]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of female participants with a categorical change in pleasure subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.412, Chi-squared — [p-value comment as in outcome 25, analysis 10]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 12: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of female participants with a categorical change in pleasure subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.030, Chi-squared — [p-value comment as in outcome 25, analysis 10]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 13: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of male participants with a categorical change in desire/frequency subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.024, Chi-squared — [p-value comment as in outcome 25, analysis 13]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 14: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of male participants with a categorical change in desire/frequency subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.250, Chi-squared — [p-value comment as in outcome 25, analysis 13]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 15: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of male participants with a categorical change in desire/frequency subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.489, Chi-squared — [p-value comment as in outcome 25, analysis 13]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 16: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of female participants with a categorical change in desire/frequency subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.682, Chi-squared — [p-value comment as in outcome 25, analysis 16]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 17: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of female participants with a categorical change in desire/frequency subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.953, Chi-squared — [p-value comment as in outcome 25, analysis 16]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 18: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of female participants with a categorical change in desire/frequency subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.803, Chi-squared — [p-value comment as in outcome 25, analysis 16]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 19: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of male participants with a categorical change in desire/interest subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.694, Chi-squared — [p-value comment as in outcome 25, analysis 19]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 20: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of male participants with a categorical change in desire/interest subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.835, Chi-squared — [p-value comment as in outcome 25, analysis 19]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 21: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of male participants with a categorical change in desire/interest subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.435, Chi-squared — [p-value comment as in outcome 25, analysis 19]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 22: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of female participants with a categorical change in desire/interest subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.379, Chi-squared — [p-value comment as in outcome 25, analysis 22]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 23: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of female participants with a categorical change in desire/interest subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.247, Chi-squared — [p-value comment as in outcome 25, analysis 22]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 24: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of female participants with a categorical change in desire/interest subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.784, Chi-squared — [p-value comment as in outcome 25, analysis 22]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 25: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of male participants with a categorical change in arousal subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.696, Chi-squared — [p-value comment as in outcome 25, analysis 25]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 26: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of male participants with a categorical change in arousal subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.725, Chi-squared — [p-value comment as in outcome 25, analysis 25]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 27: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of male participants with a categorical change in arousal subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.899, Chi-squared — [p-value comment as in outcome 25, analysis 25]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 28: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of female participants with a categorical change in arousal subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.782, Chi-squared — [p-value comment as in outcome 25, analysis 28]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 29: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of female participants with a categorical change in arousal subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.307, Chi-squared — [p-value comment as in outcome 25, analysis 28]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 30: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of female participants with a categorical change in arousal subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.457, Chi-squared — [p-value comment as in outcome 25, analysis 28]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 31: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of male participants with a categorical change in orgasm subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.712, Chi-squared — [p-value comment as in outcome 25, analysis 31]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 32: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of male participants with a categorical change in orgasm subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.403, Chi-squared — [p-value comment as in outcome 25, analysis 31]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 33: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of male participants with a categorical change in orgasm subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.713, Chi-squared — [p-value comment as in outcome 25, analysis 31]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 34: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of female participants with a categorical change in orgasm subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.498, Chi-squared — [p-value comment as in outcome 25, analysis 34]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 35: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of female participants with a categorical change in orgasm subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.963, Chi-squared — [p-value comment as in outcome 25, analysis 34]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 36: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of female participants with a categorical change in orgasm subscore from baseline to 12 weeks in the Sexual Functioning Questionnaire (CSFQ); Test type: Superiority or Other; p = 0.338, Chi-squared — [p-value comment as in outcome 25, analysis 34]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test

27. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Portland Neurotoxicity Scale - Total Score and Subscale Scores
Description: The Portland Neurotoxicity Scale is a 15-item, patient-completed questionnaire designed to assess the degree of impact of anti-epileptic drug therapy on a number of cognitive and somatomotor parameters. The total score ranges from 15-135 with higher scores indicating more toxicity. The cognitive toxicity score ranges from 10-90 and the somatomotor toxicity score ranges from 5-45, for both higher scores indicate more toxicity. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 126 | 129 | 129
units on a scale
  total, n=122, n=126, n=128 | -6.27 (1.63) | -8.92 (1.70) | -7.29 (1.59)
  cognitive toxicity, n=126, n=129, n=128 | -5.12 (1.18) | -6.23 (1.23) | -5.29 (1.16)
  somatomotor toxicity, n=122, n=126, n=129 | -1.36 (0.51) | -2.58 (0.54) | -1.91 (0.50)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Scale Total Score; Test type: Superiority or Other; p = 0.645, Mixed Models Analysis — P-value is for total. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Scale Total Score; Test type: Superiority or Other; p = 0.248, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Scale Total Score; Test type: Superiority or Other; p = 0.470, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Cognitive Toxicity Score; Test type: Superiority or Other; p = 0.914, Mixed Models Analysis — P-value is for cognitive toxicity. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Cognitive Toxicity Score; Test type: Superiority or Other; p = 0.505, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 4]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Cognitive Toxicity Score; Test type: Superiority or Other; p = 0.570, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 4]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Scale Somatomotor Toxicity Score; Test type: Superiority or Other; p = 0.430, Mixed Models Analysis — P-value is for somatomotor toxicity. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Scale Somatomotor Toxicity Score; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 7]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Portland Neurotoxicity Scale Somatomotor Toxicity Score; Test type: Superiority or Other; p = 0.341, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 7]; [statistical method as in outcome 3, analysis 1]

28. Secondary Outcome: Categorial Change From Baseline to 12 Weeks in Portland Neurotoxicity Scale - Total Score and Subscale Scores
Description: The Portland Neurotoxicity Scale is a 15-item, patient-completed questionnaire designed to assess the degree of impact of anti-epileptic drug therapy on a number of cognitive and somatomotor parameters. Categories: better=negative change in score; same=no change in score; worse=positive change in score.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 126 | 129 | 129
participants
  better, total; n=122, n=126, n=128 | 68 | 84 | 86
  same, total; n=122, n=126, n=128 | 8 | 5 | 4
  worse, total; n=122, n=126, n=128 | 46 | 37 | 38
  better, cognitive toxicity; n=126, n=129, n=128 | 75 | 80 | 82
  same, cognitive toxicity; n=126, n=129, n=128 | 9 | 6 | 5
  worse, cognitive toxicity; n=126, n=129, n=128 | 42 | 43 | 41
  better, somatomotor toxicity; n=122, n=126, n=129 | 60 | 74 | 74
  same, somatomotor toxicity; n=122, n=126, n=129 | 15 | 19 | 19
  worse, somatomotor toxicity; n=122, n=126, n=129 | 47 | 33 | 36
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale total score; Test type: Superiority or Other; p = 0.130, Chi-squared — [p-value comment as in outcome 23, analysis 1]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale total score; Test type: Superiority or Other; p = 0.192, Chi-squared — [p-value comment as in outcome 23, analysis 1]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale total score; Test type: Superiority or Other; p = 0.936, Chi-squared — [p-value comment as in outcome 23, analysis 1]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale cognitive toxicity score; Test type: Superiority or Other; p = 0.480, Chi-squared — P-value is for cognitive toxicity. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale cognitive toxicity score; Test type: Superiority or Other; p = 0.690, Chi-squared — [p-value comment as in outcome 28, analysis 4]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale cognitive toxicity score; Test type: Superiority or Other; p = 0.923, Chi-squared — [p-value comment as in outcome 28, analysis 4]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale somatomotor toxicity score; Test type: Superiority or Other; p = 0.202, Chi-squared — P-value is for somatomotor toxicity. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale somatomotor toxicity score; Test type: Superiority or Other; p = 0.114, Chi-squared — [p-value comment as in outcome 28, analysis 7]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with a categorial change from baseline to 12 weeks in the Portland Neurotoxicity Scale somatomotor toxicity score; Test type: Superiority or Other; p = 0.954, Chi-squared — [p-value comment as in outcome 28, analysis 7]; Pairwise p-values come from the Likelihood-Ratio Chi-squared test

29. Secondary Outcome: Path Analysis of Improvement in Pain Through Improvement in Depressive Symptoms
Description: Contribution to reduction in pain directly by treatment and indirectly by treatment through the reduction of depressive symptoms using path analysis. The direct treatment effect estimates the mean drug difference in pain reduction directly through treatment; the indirect treatment effect estimates the contribution that treatment plays to the mean drug difference in pain reduction indirectly through the reduction in mood symptoms; the total effect estimates the drug difference in reducing pain in sum through the specified path of direct and indirect treatment effects.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Number; unit: coefficient
Groups:
- Ordinary Coefficient: Beta-coefficient from regression analyses estimating direct and indirect treatment effects expressed in the observed scale of measurement of the dependent variable.
Arm/Group | Ordinary Coefficient
Number analyzed (Participants) | 234
coefficient
  Direct Treatment Effect | -0.449
  Indirect Treatment Effect | 0.014
  Total Treatment Effect | -0.435
Statistical Analysis 1: Comparison: Ordinary Coefficient; Test type: Superiority or Other; p = 0.107, Regression, Linear — P-value for Direct Treatment Effect. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for tests of direct and indirect effects

30. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Beck Depression Inventory II (BDI-II) Total Score
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 121 | 125 | 125
units on a scale | -2.57 (0.58) | -3.13 (0.60) | -2.54 (0.57)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BDI-II total score; Test type: Superiority or Other; p = 0.968, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in BDI-II total score; Test type: Superiority or Other; p = 0.492, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in BDI-II total score; Test type: Superiority or Other; p = 0.463, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

31. Secondary Outcome: Categorical Change From Baseline to 12 Weeks in Number of Patients Using Health Care as Measured by the Resource Utilization Scale
Description: The Resource Utilization Scale measures direct and indirect costs (collected only for US sites). Direct costs include inpatient and outpatient costs, while indirect costs include lost days of work and caregiver time spent with patients. Inpatient costs include costs associated with hospitalizations and time spent in emergency rooms and psychiatric rooms. Outpatient costs include costs associated with visits to various health care providers, home health care by health care providers, and partial care.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 134 | 138 | 135
participants
  hours worked, greater, n=86, n=90, n=83 | 10 | 12 | 13
  hours worked, same, n=86, n=90, n=83 | 65 | 66 | 59
  hours worked, lower, n=86, n=90, n=83 | 11 | 12 | 11
  hours volunteered, greater, n=86, n=91, n=82 | 7 | 8 | 10
  hours volunteered, same, n=86, n=91, n=82 | 66 | 77 | 66
  hours volunteered, lower, n=86, n=91, n=82 | 13 | 6 | 6
  psychiatric visits, greater, n=92, n=93, n=90 | 2 | 0 | 2
  psychiatric visits, same, n=92, n=93, n=90 | 88 | 91 | 84
  psychiatric visits, lower, n=92, n=93, n=90 | 2 | 2 | 4
  outpatient group visits, greater, n=91, n=92, n=91 | 0 | 0 | 1
  outpatient group visits, same, n=91, n=92, n=91 | 90 | 92 | 89
  outpatient group visits, lower, n=91, n=92, n=91 | 1 | 0 | 1
  outpatient ind. visits, greater, n=91, n=88, n=90 | 3 | 1 | 4
  outpatient ind. visits, same, n=91, n=88, n=90 | 84 | 84 | 81
  outpatient ind. visits, lower, n=91, n=88, n=90 | 4 | 3 | 5
  days of partial care, greater, n=93, n=95, n=90 | 2 | 1 | 2
  days of partial care, same, n=93, n=95, n=90 | 91 | 94 | 87
  days of partial care, lower, n=93, n=95, n=90 | 0 | 0 | 1
  nights of partial care, greater, n=92, n=95, n=91 | 1 | 1 | 2
  nights of partial care, same, n=92, n=95, n=91 | 91 | 94 | 89
  nights of partial care, lower, n=92, n=95, n=91 | 0 | 0 | 0
  ER visits-psychiatric, greater, n=93, n=94, n=91 | 0 | 0 | 0
  ER visits-psychiatric, same, n=93, n=94, n=91 | 91 | 94 | 91
  ER visits-psychiatric, lower, n=93, n=94, n=91 | 2 | 0 | 0
  ER visits-nonpsychiatric, greater,n=91, n=95, n=88 | 3 | 4 | 4
  ER visits-nonpsychiatric, same,n=91, n=95, n=88 | 83 | 85 | 78
  ER visits-nonpsychiatric, lower,n=91, n=95, n=88 | 5 | 6 | 6
  phone mental health, greater,n=94, n=95, n=90 | 1 | 1 | 2
  phone mental health, same,n=94, n=95, n=90 | 92 | 93 | 87
  phone mental health, lower,n=94, n=95, n=90 | 1 | 1 | 1
  nonpsychiatric visits, greater, n=89, n=94, n=83 | 24 | 20 | 18
  nonpsychiatric visits, same, n=89, n=94, n=83 | 44 | 46 | 45
  nonpsychiatric visits, lower, n=89, n=94, n=83 | 21 | 28 | 20
  unpaid care, greater, n=84, n=87, n=86 | 2 | 0 | 0
  unpaid care, same, n=84, n=87, n=86 | 82 | 87 | 85
  unpaid care, lower, n=84, n=87, n=86 | 0 | 0 | 1
  missed work caregiver, greater, n=6, n=9, n=5 | 0 | 0 | 0
  missed work caregiver, same, n=6, n=9, n=5 | 6 | 8 | 5
  missed work caregiver, lower, n=6, n=9, n=5 | 0 | 1 | 0
  paid care, greater, n=60, n=58, n=58 | 0 | 0 | 0
  paid care, same, n=60, n=58, n=58 | 60 | 58 | 58
  paid care, less, n=60, n=58, n=58 | 0 | 0 | 0

32. Secondary Outcome: Summary of Number of Participants Who Discontinued
Description: Number of participants who discontinued. The reasons for discontinuation are presented in the participant flow.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 134 | 138 | 135
participants | 38 | 51 | 36

33. Secondary Outcome: Time to First ≥ 30% Reduction in Weekly Mean 24 Hour Average Pain Score
Description: This is the number of days required to first achieve a nominal outcome reflecting whether or not a clinically-important efficacy outcome was achieved. It is based on a comparison between baseline and post-baseline scores on an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Used were the weekly mean of the scores of the average pain severity over the last 24 hours. The weekly averages were based on daily assessments recorded by patients in their diaries.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
days | 35.0 [28.0 to 55.0] | 28.0 [20.0 to 35.0] | 28.0 [21.0 to 35.0]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in time to first ≥ 30% reduction in weekly mean 24 hour average pain score; Test type: Superiority or Other; p = 0.103, Log Rank — [p-value comment as in outcome 5, analysis 1]; Pairwise p-values come from the log-rank test comparing treatment-specific time-to-event curves constructed using the Kaplan-Meier technique
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in time to first ≥ 30% reduction in weekly mean 24 hour average pain score; Test type: Superiority or Other; p = 0.167, Log Rank — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in time to first ≥ 30% reduction in weekly mean 24 hour average pain score; Test type: Superiority or Other; p = 0.919, Log Rank — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 33, analysis 1]

34. Secondary Outcome: Time to First ≥ 50 % Reduction in Weekly Mean 24 Hour Average Pain Score
Description: This is the number of days to first achieve ≥50% reduction, baseline to endpoint, in the weekly means of the 24-hour average pain severity via daily patient assessments using an ordinal scale (scores from 0 (no pain) to 10 (worst possible pain). The median time to first ≥50% reduction with some measure of dispersion could not be calculated for each treatment group. The number of patients who reached a ≥50% reduction in weekly mean 24 hour average pain score are presented in outcome measure 20.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Time to First Sustained Response in Weekly Mean 24 Hour Average Pain Score
Description: This is the number of days to first achieve an outcome using the weekly means of the 24-hour average pain severity via daily patient assessments using an ordinal scale (scores from 0 (no pain) to 10 (worst possible pain). Sustained response: ≥30% reduction, baseline to endpoint, with 30% reduction from baseline ≥2 weeks prior to endpoint, remaining at ≥20% reduction between. The median time to sustained response with some measure of dispersion could not be calculated for each treatment group.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 0 | 0 | 0

36. Secondary Outcome: Time to First ≥ 2 Points Reduction in Weekly Mean 24 Hour Average Pain Score
Description: as for outcome 33
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 127 | 120 | 125
days | 56.0 [39.0 to 80.0] | 35.0 [28.0 to 53.0] | 28.0 [22.0 to 42.0]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in time to first ≥ 2 points reduction in weekly mean 24 hour average pain score; Test type: Superiority or Other; p = 0.008, Log Rank — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 33, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in time to first ≥ 2 points reduction in weekly mean 24 hour average pain score; Test type: Superiority or Other; p = 0.033, Log Rank — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 33, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in time to first ≥ 2 points reduction in weekly mean 24 hour average pain score; Test type: Superiority or Other; p = 0.688, Log Rank — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 33, analysis 1]

37. Secondary Outcome: Weekly Mean Change in 24 Hour Average Pain Severity +/- Generalized Anxiety Disorder (GAD)
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the average pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries.
  It was planned to analyze participants stratified by the presence or absence of a co-morbidity with GAD. However, due to the low number of participants with GAD in the study this analysis was not possible.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Weekly Mean Change From Baseline to 12 Weeks in 24 Hour Average Pain Severity - Only Participants Who Adhered to Key Protocol Requirements (Per-Protocol Population)
Description: Ordinal scale: 0=no pain, 10=worst possible pain. Data=weekly mean of scores of average pain severity over last 24 hours (h). Scores: daily assessments recorded by patients in diaries. Only patients adhering to key protocol criteria included: baseline Weekly Mean 24h Average Pain Score ≥4; 80-120% compliant with study Drug, each visit; baseline Michigan Neuropathy Screening Instrument Physical Assessment Total Score ≥3; gabapentin taper ≤14 days, no HbA1c ≥12% post randomization; no contraindicated medications used. Least-squares means=adjustment due to baseline severity + investigative site.
Time Frame: baseline, 12 weeks
Population: The per-protocol sub-population of all randomized participants with a baseline value and >= 1 non-missing post-baseline value (modified intent-to-treat population) was included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 94 | 77 | 103
units on a scale
  baseline | 5.74 (1.30) | 6.02 (1.60) | 5.74 (1.42)
  change | -2.12 (0.23) | -2.58 (0.27) | -2.40 (0.23)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Weekly mean change from baseline to 12 weeks in 24 hour average pain severity score when analyzing only treatment-compliant participants; Test type: Superiority or Other; p = 0.365, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Change=Treatment+InvestigatorGroup+Week+Baseline+Treatment*Week+Baseline*Week with participant is as a random effect, Kenward-Roger approximation; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.33 to 0.90]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in Weekly mean change from baseline to 12 weeks in 24 hour average pain severity score when analyzing only treatment-compliant participants; Test type: Superiority or Other; p = 0.172, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 38, analysis 1]; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.20 to 1.13]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in Weekly mean change from baseline to 12 weeks in 24 hour average pain severity score when analyzing only treatment-compliant participants; Test type: Superiority or Other; p = 0.594, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 38, analysis 1]; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.49 to 0.85]

39. Secondary Outcome: Weekly Mean Change in 24 Hour Average Pain Severity by Week by Gabapentin Exposure Subgroup (de Novo Versus Prior Use)
Description: This is an ordinal scale with scores from 0 (no pain) to 10 (worst possible pain). Data presented represent the weekly mean of the scores of the average pain severity over the last 24 hours. Scores are based on daily assessments recorded by patients in their diaries. De novo: use of gabapentin for <56 contiguous days prior to randomization. Prior use: use of gabapentin for >=56 contiguous days prior to randomization. Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks, 9 weeks, 10 weeks, 11 weeks, 12 weeks
Population: Analyzed were all participants with a baseline and at least 1 non-missing post-baseline value. Last observation carried forward analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 134 | 138 | 135
units on a scale
  de novo, baseline | 5.24 (1.07) | 5.39 (1.48) | 5.49 (1.45)
  de novo, week 1 | -0.22 (0.24) | -0.71 (0.27) | -0.38 (0.25)
  de novo, week 2 | -0.39 (0.27) | -1.22 (0.31) | -1.10 (0.28)
  de novo, week 3 | -0.71 (0.30) | -1.83 (0.30) | -1.62 (0.30)
  de novo, week 4 | -0.84 (0.32) | -2.35 (0.35) | -1.67 (0.32)
  de novo, week 5 | -0.95 (0.33) | -2.65 (0.37) | -1.81 (0.33)
  de novo, week 6 | -1.09 (0.34) | -2.64 (0.38) | -1.88 (0.34)
  de novo, week 7 | -1.08 (0.34) | -2.73 (0.38) | -2.07 (0.34)
  de novo, week 8 | -1.26 (0.35) | -2.78 (0.39) | -2.06 (0.35)
  de novo, week 9 | -1.21 (0.34) | -2.89 (0.38) | -2.10 (0.35)
  de novo, week 10 | -1.42 (0.35) | -2.86 (0.39) | -1.92 (0.35)
  de novo, week 11 | -1.48 (0.35) | -2.98 (0.39) | -2.09 (0.35)
  de novo, week 12 | -1.62 (0.36) | -3.08 (0.40) | -2.10 (0.36)
  prior use, baseline | 5.91 (1.55) | 5.99 (1.52) | 5.92 (1.48)
  prior use, week 1 | -0.30 (0.17) | -0.48 (0.16) | -0.65 (0.17)
  prior use, week 2 | -0.70 (0.19) | -0.99 (0.19) | -1.28 (0.19)
  prior use, week 3 | -1.18 (0.20) | -1.32 (0.20) | -1.68 (0.21)
  prior use, week 4 | -1.64 (0.21) | -1.61 (0.22) | -1.75 (0.22)
  prior use, week 5 | -1.72 (0.22) | -1.95 (0.23) | -1.96 (0.22)
  prior use, week 6 | -1.92 (0.23) | -2.03 (0.23) | -1.98 (0.23)
  prior use, week 7 | -1.93 (0.23) | -2.14 (0.23) | -2.17 (0.23)
  prior use, week 8 | -1.89 (0.23) | -2.16 (0.24) | -2.31 (0.23)
  prior use, week 9 | -2.04 (0.23) | -2.38 (0.24) | -2.37 (0.23)
  prior use, week 10 | -2.14 (0.23) | -2.45 (0.24) | -2.44 (0.24)
  prior use, week 11 | -2.27 (0.23) | -2.46 (0.24) | -2.41 (0.24)
  prior use, week 12 | -2.39 (0.23) | -2.46 (0.24) | -2.53 (0.24)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 1; Test type: Superiority or Other; p = 0.622, Mixed Models Analysis — P-value is for de novo, week 1. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; Model Change=Investigator+ Treatment+Week+Subgroup+Baseline+Treatment*Week+ Baseline*Week+Subgroup*Week+Subgroup*Treatment+Subgroup*Treatment*Week; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.48 to 0.80]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 1; Test type: Superiority or Other; p = 0.153, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 1]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.18 to 1.16]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 1; Test type: Superiority or Other; p = 0.344, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 1]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.35 to 1.00]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 2; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis — P-value is for de novo, week 2. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-0.02 to 1.45]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 2; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 4]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.07 to 1.59]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 2; Test type: Superiority or Other; p = 0.762, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 4]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.66 to 0.90]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 3; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis — P-value is for de novo, week 3. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [0.09 to 1.73]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 3; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — P-value is for de nove, 3 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [0.27 to 1.97]
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 3; Test type: Superiority or Other; p = 0.619, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 8]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.63 to 1.06]
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 4; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis — P-value is for de novo, 4 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.03 to 1.69]
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 4; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 10]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [0.61 to 2.41]
Statistical Analysis 12: Comparison: Duloxetine vs Gabapentin + Duloxetine; [analysis description as in outcome 39, analysis 3]; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis — P-value is for de nove, 4 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-0.23 to 1.58]
Statistical Analysis 13: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 5; Test type: Superiority or Other; p = 0.065, Mixed Models Analysis — P-value is for de novo, 5 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.05 to 1.76]
Statistical Analysis 14: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 5; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 13]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.70, 95% CI 2-sided [0.75 to 2.65]
Statistical Analysis 15: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 5; Test type: Superiority or Other; p = 0.079, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 13]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.10 to 1.79]
Statistical Analysis 16: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 6; Test type: Superiority or Other; p = 0.093, Mixed Models Analysis — P-value is for de novo, 6 week. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.13 to 1.71]
Statistical Analysis 17: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 6; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — P-value is for de novo, 6 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.56, 95% CI 2-sided [0.59 to 2.53]
Statistical Analysis 18: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 6; Test type: Superiority or Other; p = 0.119, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 17]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-0.20 to 1.74]
Statistical Analysis 19: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 7; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — P-value is for de novo, 7 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [0.06 to 1.91]
Statistical Analysis 20: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 7; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 19]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.65, 95% CI 2-sided [0.68 to 2.61]
Statistical Analysis 21: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 7; Test type: Superiority or Other; p = 0.178, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 19]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-0.30 to 1.63]
Statistical Analysis 22: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 8; Test type: Superiority or Other; p = 0.093, Mixed Models Analysis — P-value is for de novo, 8 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.14 to 1.75]
Statistical Analysis 23: Comparison: Pregabalin vs Duloxetine; [analysis description as in outcome 39, analysis 20]; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 22]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.52, 95% CI 2-sided [0.53 to 2.51]
Statistical Analysis 24: Comparison: Duloxetine vs Gabapentin + Duloxetine; [analysis description as in outcome 39, analysis 3]; Test type: Superiority or Other; p = 0.157, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 22]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-0.28 to 1.71]
Statistical Analysis 25: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 9; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis — P-value is for de novo, 9 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-0.05 to 1.82]
Statistical Analysis 26: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 9; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 25]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [0.70 to 2.66]
Statistical Analysis 27: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 9; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 25]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.19 to 1.77]
Statistical Analysis 28: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 10; Test type: Superiority or Other; p = 0.295, Mixed Models Analysis — P-value is for de novo, 10 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.44 to 1.46]
Statistical Analysis 29: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 10; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 28]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [0.45 to 2.44]
Statistical Analysis 30: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 10; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 28]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.06 to 1.94]
Statistical Analysis 31: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 11; Test type: Superiority or Other; p = 0.208, Mixed Models Analysis — P-value is for de novo, 11 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.35 to 1.58]
Statistical Analysis 32: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 11; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 31]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [0.49 to 2.51]
Statistical Analysis 33: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 11; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 31]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-0.13 to 1.89]
Statistical Analysis 34: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 12; Test type: Superiority or Other; p = 0.328, Mixed Models Analysis — P-value is for de novo, 12 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-0.49 to 1.45]
Statistical Analysis 35: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 12; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 34]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [0.44 to 2.47]
Statistical Analysis 36: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin de novo group in change in 24 hour average pain severity at Week 12; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 34]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [-0.04 to 1.99]
Statistical Analysis 37: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 1; Test type: Superiority or Other; p = 0.117, Mixed Models Analysis — P-value is for prior use, 1 week. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.09 to 0.79]
Statistical Analysis 38: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 1; Test type: Superiority or Other; p = 0.412, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 37]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.25 to 0.62]
Statistical Analysis 39: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 1; Test type: Superiority or Other; p = 0.445, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 37]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.60 to 0.26]
Statistical Analysis 40: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 2; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — P-value is for prior use, 2 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.07 to 1.09]
Statistical Analysis 41: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 2; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 40]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.21 to 0.79]
Statistical Analysis 42: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 2; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 40]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.79 to 0.21]
Statistical Analysis 43: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 3; Test type: Superiority or Other; p = 0.075, Mixed Models Analysis — P-value is for prior use, 3 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.05 to 1.04]
Statistical Analysis 44: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 3; Test type: Superiority or Other; p = 0.634, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 43]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.42 to 0.68]
Statistical Analysis 45: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 3; Test type: Superiority or Other; p = 0.193, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 43]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.91 to 0.19]
Statistical Analysis 46: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 4; Test type: Superiority or Other; p = 0.688, Mixed Models Analysis — P-value is for prior use, 4 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.46 to 0.70]
Statistical Analysis 47: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 4; Test type: Superiority or Other; p = 0.944, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 46]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.60 to 0.56]
Statistical Analysis 48: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 4; Test type: Superiority or Other; p = 0.640, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 46]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.73 to 0.45]
Statistical Analysis 49: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 5; Test type: Superiority or Other; p = 0.439, Mixed Models Analysis — P-value is for prior use, 5 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.37 to 0.84]
Statistical Analysis 50: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 5; Test type: Superiority or Other; p = 0.461, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 49]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.38 to 0.84]
Statistical Analysis 51: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 5; Test type: Superiority or Other; p = 0.976, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 49]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.62 to 0.60]
Statistical Analysis 52: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 6; Test type: Superiority or Other; p = 0.829, Mixed Models Analysis — P-value is for prior use, 6 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.55 to 0.68]
Statistical Analysis 53: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 6; Test type: Superiority or Other; p = 0.713, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 52]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.50 to 0.74]
Statistical Analysis 54: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 6; Test type: Superiority or Other; p = 0.878, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 52]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.58 to 0.67]
Statistical Analysis 55: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 7; Test type: Superiority or Other; p = 0.447, Mixed Models Analysis — P-value is for prior use, 7 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.38 to 0.85]
Statistical Analysis 56: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 7; Test type: Superiority or Other; p = 0.511, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 55]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.41 to 0.83]
Statistical Analysis 57: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 7; Test type: Superiority or Other; p = 0.924, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 55]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.65 to 0.59]
Statistical Analysis 58: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 8; Test type: Superiority or Other; p = 0.185, Mixed Models Analysis — P-value is for prior use, 8 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.20 to 1.06]
Statistical Analysis 59: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 8; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 58]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.37 to 0.91]
Statistical Analysis 60: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 8; Test type: Superiority or Other; p = 0.636, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 58]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.79 to 0.49]
Statistical Analysis 61: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 9; Test type: Superiority or Other; p = 0.304, Mixed Models Analysis — P-value is for prior use, 9 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.30 to 0.95]
Statistical Analysis 62: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 9; Test type: Superiority or Other; p = 0.295, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 61]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.29 to 0.97]
Statistical Analysis 63: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 9; Test type: Superiority or Other; p = 0.975, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 61]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.62 to 0.64]
Statistical Analysis 64: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 10; Test type: Superiority or Other; p = 0.349, Mixed Models Analysis — P-value is for prior use, 10 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.33 to 0.93]
Statistical Analysis 65: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 10; Test type: Superiority or Other; p = 0.351, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 64]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.34 to 0.94]
Statistical Analysis 66: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 10; Test type: Superiority or Other; p = 0.992, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 64]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.64 to 0.65]
Statistical Analysis 67: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 11; Test type: Superiority or Other; p = 0.681, Mixed Models Analysis — P-value is for prior use, 11 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.50 to 0.77]
Statistical Analysis 68: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 11; Test type: Superiority or Other; p = 0.569, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 67]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.46 to 0.83]
Statistical Analysis 69: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 11; Test type: Superiority or Other; p = 0.871, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 67]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.60 to 0.70]
Statistical Analysis 70: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 12; Test type: Superiority or Other; p = 0.675, Mixed Models Analysis — P-value is for prior use, 12 weeks. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.50 to 0.78]
Statistical Analysis 71: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 12; Test type: Superiority or Other; p = 0.823, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 70]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.57 to 0.72]
Statistical Analysis 72: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the gabapentin prior use group in change in 24 hour average pain severity at Week 12; Test type: Superiority or Other; p = 0.850, Mixed Models Analysis — [p-value comment as in outcome 39, analysis 70]; [statistical method as in outcome 39, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.72 to 0.59]

40. Secondary Outcome: Discontinuations for Abnormal Laboratory Analytes, Vital Signs, Overall and for Each Measure
Description: Presented are numbers of participants who discontinued due to a change from baseline in laboratory analytes or vital signs.
Time Frame: baseline through 12 weeks
Population: All randomized patients.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 134 | 138 | 135
participants
  Increased blood creatinine | 0 | 0 | 1
  Increased blood glucose | 1 | 0 | 0

41. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Blood Pressure
Description: Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeter mercury
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 130 | 133 | 132
millimeter mercury
  Diastolic | 0.18 (0.92) | 2.24 (0.97) | -0.79 (0.91)
  Systolic | -3.31 (1.44) | -3.08 (1.54) | -2.08 (1.43)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in diastolic blood pressure; Test type: Superiority or Other; p = 0.448, Mixed Models Analysis — P-value is for diastolic. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in diastolic blood pressure; Test type: Superiority or Other; p = 0.118, Mixed Models Analysis — [p-value comment as in outcome 41, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in diastolic blood pressure; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — [p-value comment as in outcome 41, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in systolic blood pressure; Test type: Superiority or Other; p = 0.537, Mixed Models Analysis — P-value is for systolic. P-values are not adjusted for multiple comparisons. The a priori significance level was set to 0.05 for treatment comparisons and 0.10 for tests of interaction; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in systolic blood pressure; Test type: Superiority or Other; p = 0.911, Mixed Models Analysis — [p-value comment as in outcome 41, analysis 4]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in systolic blood pressure; Test type: Superiority or Other; p = 0.627, Mixed Models Analysis — [p-value comment as in outcome 41, analysis 4]; [statistical method as in outcome 3, analysis 1]

42. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Heart Rate
Description: Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 130 | 133 | 132
beats per minute | -1.30 (0.97) | 0.80 (1.02) | 1.05 (0.96)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in heart rate; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in heart rate; Test type: Superiority or Other; p = 0.130, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in heart rate; Test type: Superiority or Other; p = 0.850, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

43. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Body Weight
Description: Least-squares means represent adjustment due to baseline severity and investigative site.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 130 | 132 | 132
kilogram | 1.00 (0.36) | -2.39 (0.38) | -1.06 (0.36)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in body weight; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in body weight; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in body weight; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]

44. Secondary Outcome: Number of Participants With Treatment-emergent Elevated Blood Pressure
Description: Elevated systolic blood pressure: >=130 millimeter mercury (mm Hg) + an increase of >=10 mm Hg if baseline <130 mm Hg.
  Elevated diastolic blood pressure: >=85 mm Hg + an increase of >=10 mm Hg if baseline <85 mm Hg.
Time Frame: baseline through 12 weeks
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 94 | 98 | 100
participants
  diastolic, n=94, n=98, n=100 | 11 | 12 | 13
  systolic, n=42, n=39, n=56 | 20 | 15 | 16
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in the number of participants with elevated diastolic blood pressure; Test type: Superiority or Other; p = 0.830, Fisher Exact — P-value is for diastolic. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in the number of participants with elevated diastolic blood pressure; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 44, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in the number of participants with elevated diastolic blood pressure; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 44, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in the number of participants with elevated systolic blood pressure; Test type: Superiority or Other; p = 0.060, Fisher Exact — P-value is for systolic. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in the number of participants with elevated systolic blood pressure; Test type: Superiority or Other; p = 0.502, Fisher Exact — [p-value comment as in outcome 44, analysis 4]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; [analysis description as in outcome 44, analysis 4]; Test type: Superiority or Other; p = 0.376, Fisher Exact — [p-value comment as in outcome 44, analysis 4]

45. Secondary Outcome: Number of Participants With Treatment-Emergent Elevated Heart Rate
Description: Elevated heart rate: >=100 beats per minute (bpm) + an increase of >=10 bpm if baseline <100 bpm.
Time Frame: baseline through 12 weeks
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 126 | 128 | 127
participants | 2 | 9 | 6
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated heart rate; Test type: Superiority or Other; p = 0.281, Fisher Exact — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated heart rate; Test type: Superiority or Other; p = 0.060, Fisher Exact — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated heart rate; Test type: Superiority or Other; p = 0.596, Fisher Exact — [p-value comment as in outcome 5, analysis 1]

46. Secondary Outcome: Number of Participants With Treatment-Emergent Changes in Body Weight
Description: Treatment-emergent high body weight: weight at last visit >=107% of baseline weight.
  Treatment-emergent low body weight: weight at last visit <=93% of baseline weight.
Time Frame: baseline through 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 130 | 132 | 132
participants
  high | 6 | 1 | 3
  low | 2 | 10 | 8
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of patients with treatment-emergent high body weight; Test type: Superiority or Other; p = 0.332, Fisher Exact — P-value is for high. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of patients with treatment-emergent high body weight; Test type: Superiority or Other; p = 0.065, Fisher Exact — [p-value comment as in outcome 46, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of patients with treatment-emergent high body weight; Test type: Superiority or Other; p = 0.622, Fisher Exact — [p-value comment as in outcome 46, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of patients with treatment-emergent low body weight; Test type: Superiority or Other; p = 0.103, Fisher Exact — P-value is for low. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of patients with treatment-emergent low body weight; Test type: Superiority or Other; p = 0.034, Fisher Exact — [p-value comment as in outcome 46, analysis 4]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of patients with treatment-emergent low body weight; Test type: Superiority or Other; p = 0.808, Fisher Exact — [p-value comment as in outcome 46, analysis 4]

47. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Hepatic Enzyme Serum Levels
Description: Aspartate aminotransferase = AST Alanine aminotransferase = ALT Gamma glutamyl transferase = GGT Alkaline phosphatase = AlkPhos
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 121 | 123 | 120
units/liter
  baseline, AST, n=119, n=121, n=118 | 22.55 (7.64) | 22.84 (8.70) | 23.42 (8.19)
  change, AST, n=119, n=121, n=118 | 1.12 (7.62) | -0.52 (6.82) | -0.48 (7.71)
  baseline, ALT, n=120, n=122, n=120 | 23.88 (10.14) | 25.04 (13.18) | 24.39 (10.79)
  change, ALT, n=120, n=122, n=120 | -0.13 (7.86) | -0.16 (10.45) | 0.03 (9.53)
  baseline, GGT, n=121, n=123, n=120 | 40.80 (53.08) | 34.29 (25.53) | 43.93 (48.45)
  change, GGT, n=121, n=123, n=120 | 1.17 (39.35) | -3.03 (15.56) | -2.55 (22.85)
  baseline, AlkPhos, n=121, n=123, n=120 | 84.97 (29.36) | 83.74 (38.27) | 82.18 (28.39)
  change, AlkPhos, n=121, n=123, n=120 | 2.80 (40.32) | 0.55 (18.21) | 1.78 (12.84)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 in AST; Test type: Superiority or Other; p = 0.055, t-test, 2 sided — P-value is for AST. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; Analysis of Variance model & t-test: Rank-transformed Change=InvestigatorGroup+Treatment. Last-observation-carried-forward imputation was implemented
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 in AST; Test type: Superiority or Other; p = 0.051, t-test, 2 sided — [p-value comment as in outcome 47, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; [analysis description as in outcome 47, analysis 1]; Test type: Superiority or Other; p = 0.993, t-test, 2 sided — [p-value comment as in outcome 47, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 in ALT; Test type: Superiority or Other; p = 0.928, t-test, 2 sided — P-value is for ALT. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 in ALT; Test type: Superiority or Other; p = 0.609, t-test, 2 sided — [p-value comment as in outcome 47, analysis 4]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 in ALT; Test type: Superiority or Other; p = 0.675, t-test, 2 sided — [p-value comment as in outcome 47, analysis 4]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 in GGT; Test type: Superiority or Other; p = 0.985, t-test, 2 sided — P-value is for GGT. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 in GGT; Test type: Superiority or Other; p = 0.847, t-test, 2 sided — [p-value comment as in outcome 47, analysis 7]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 9: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 in GGT; Test type: Superiority or Other; p = 0.832, t-test, 2 sided — [p-value comment as in outcome 47, analysis 7]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 in AlkPhos; Test type: Superiority or Other; p = 0.169, t-test, 2 sided — P-value is for AlkPhos. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 11: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 in AlkPhos; Test type: Superiority or Other; p = 0.910, t-test, 2 sided — [p-value comment as in outcome 47, analysis 10]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 12: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 in AlkPhos; Test type: Superiority or Other; p = 0.134, t-test, 2 sided — [p-value comment as in outcome 47, analysis 10]; [statistical method as in outcome 47, analysis 1]

48. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Total Bilirubin
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromole/liter
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 120 | 123 | 120
micromole/liter
  baseline | 8.43 (4.50) | 8.07 (3.99) | 8.23 (5.07)
  change | -0.51 (3.48) | -0.28 (2.60) | -0.42 (3.39)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 total bilirubin; Test type: Superiority or Other; p = 0.285, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 in total bilirubin; Test type: Superiority or Other; p = 0.505, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 in total bilirubin; Test type: Superiority or Other; p = 0.679, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]

49. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Fasting Plasma Glucose
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimole/liter
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 86 | 82 | 78
millimole/liter
  baseline | 8.24 (3.31) | 8.45 (3.65) | 7.99 (3.82)
  change | 0.16 (3.97) | 0.19 (2.86) | 0.67 (2.75)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in fasting blood glucose; Test type: Superiority or Other; p = 0.047, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in fasting blood glucose; Test type: Superiority or Other; p = 0.232, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in fasting blood glucose; Test type: Superiority or Other; p = 0.424, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]

50. Secondary Outcome: Mean Change From Baseline to 12 Weeks in Hemoglobin A1C
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 117 | 124 | 119
percent
  baseline | 7.57 (1.61) | 7.51 (1.44) | 7.16 (1.44)
  change | -0.12 (1.00) | -0.01 (0.71) | 0.07 (0.80)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in mean change from baseline to 12 Weeks in hemoglobin A1C; Test type: Superiority or Other; p = 0.298, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in mean change from baseline to 12 Weeks in hemoglobin A1C; Test type: Superiority or Other; p = 0.987, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in mean change from baseline to 12 Weeks in hemoglobin A1C; Test type: Superiority or Other; p = 0.297, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 47, analysis 1]

51. Secondary Outcome: Number of Patients With Treatment-Emergent Elevated Laboratory Analytes
Description: Treatment-emergent: within range at baseline, out of range after baseline. Ranges in Units/Liter (U/L). Aspartate Aminotransferase (AST): female (f): >34, male (m): >36. Alanine Aminotransferase (ALT): f:<69 years (yr) >34, ≥69yr >32; m: <69yr >43, ≥69yr >35. Total Bilirubin (TBili): >21. Gamma Glutamyl Transferase (GGT): f: <59yr >49, ≥59yr >50; m: <59yr >61, ≥59yr >50. Fasting Plasma Glucose (FPG): <59yr >6.4, ≥59yr >6.7. Hemoglobin A1C (HbA1C) >6%. Alkaline Phosphatase (AlkPhos): f: 18-50yr >106, 50-70yr >123, 70-80yr >164, ≥80yr >221; m: 18-50yr >129, 50-70yr >131, 70-80yr >156, ≥80yr >187
Time Frame: baseline through 12 weeks
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Number analyzed (Participants) | 121 | 124 | 120
participants
  AST, n=113, n=116, n=109 | 4 | 6 | 4
  ALT, n=111, n=104, n=110 | 3 | 6 | 10
  TBili, n=119, n=121, n=116 | 2 | 0 | 0
  GGT, n=102, n=105, n=96 | 2 | 6 | 6
  FPG, n=33, n=30, n=36 | 7 | 11 | 18
  HbA1C, n=17, n=18, n=29 | 6 | 2 | 10
  AlkPhos, n=112, n=114, n=113 | 4 | 3 | 4
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated AST values; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 47, analysis 1]
Statistical Analysis 2: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated AST values; Test type: Superiority or Other; p = 0.749, Fisher Exact — [p-value comment as in outcome 47, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated AST values; Test type: Superiority or Other; p = 0.750, Fisher Exact — [p-value comment as in outcome 47, analysis 1]
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated ALT values; Test type: Superiority or Other; p = 0.050, Fisher Exact — [p-value comment as in outcome 47, analysis 4]
Statistical Analysis 5: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated ALT values; Test type: Superiority or Other; p = 0.320, Fisher Exact — [p-value comment as in outcome 47, analysis 4]
Statistical Analysis 6: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated ALT values; Test type: Superiority or Other; p = 0.440, Fisher Exact — [p-value comment as in outcome 47, analysis 4]
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated TBili values; Test type: Superiority or Other; p = 0.498, Fisher Exact — P-value is for TBili. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 8: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated TBili values; Test type: Superiority or Other; p = 0.245, Fisher Exact — [p-value comment as in outcome 51, analysis 7]
Statistical Analysis 9: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated GGT values; Test type: Superiority or Other; p = 0.160, Fisher Exact — [p-value comment as in outcome 47, analysis 7]
Statistical Analysis 10: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated GGT values; Test type: Superiority or Other; p = 0.280, Fisher Exact — [p-value comment as in outcome 47, analysis 7]
Statistical Analysis 11: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated GGT values; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 47, analysis 7]
Statistical Analysis 12: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated FPG values; Test type: Superiority or Other; p = 0.023, Fisher Exact — P-value is for FPG. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 13: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated FPG values; Test type: Superiority or Other; p = 0.264, Fisher Exact — [p-value comment as in outcome 51, analysis 12]
Statistical Analysis 14: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated FPG values; Test type: Superiority or Other; p = 0.325, Fisher Exact — [p-value comment as in outcome 51, analysis 12]
Statistical Analysis 15: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated HbA1C values; Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value is for HbA1C. P-values are not adjusted for multiple comparisons. The a priori level of significance was specified to be 0.05 for between-treatment-group comparisons
Statistical Analysis 16: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated HbA1C values; Test type: Superiority or Other; p = 0.121, Fisher Exact — [p-value comment as in outcome 51, analysis 15]
Statistical Analysis 17: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated HbA1C values; Test type: Superiority or Other; p = 0.095, Fisher Exact — [p-value comment as in outcome 51, analysis 15]
Statistical Analysis 18: Comparison: Pregabalin vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and gabapentin+duloxetine in the number of participants with treatment-emergent elevated AlkPhos values; Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 47, analysis 10]
Statistical Analysis 19: Comparison: Pregabalin vs Duloxetine; Tested was the null-hypothesis that there would be no difference between pregabalin and duloxetine in the number of participants with treatment-emergent elevated AlkPhos values; Test type: Superiority or Other; p = 0.720, Fisher Exact — [p-value comment as in outcome 47, analysis 10]
Statistical Analysis 20: Comparison: Duloxetine vs Gabapentin + Duloxetine; Tested was the null-hypothesis that there would be no difference between duloxetine and gabapentin+duloxetine in the number of participants with treatment-emergent elevated AlkPhos values; Test type: Superiority or Other; p = 0.722, Fisher Exact — [p-value comment as in outcome 47, analysis 10]

ADVERSE EVENTS:
Arm/Group | Pregabalin | Duloxetine | Gabapentin + Duloxetine
Serious Adverse Events (participants affected / at risk) | 6/134 | 3/138 | 5/135
Other Adverse Events (participants affected / at risk) | 87/134 | 100/138 | 88/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=134) | Duloxetine (N=138) | Gabapentin + Duloxetine (N=135)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=134) | Duloxetine (N=138) | Gabapentin + Duloxetine (N=135)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 4 (4)
Vision blurred (Eye disorders) | 4 (4) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 6 (6) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 19 (19) | 18 (18)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (6) | 6 (11)
Asthenia (General disorders) | 0 (0) | 4 (4) | 1 (1)
Fatigue (General disorders) | 7 (7) | 16 (16) | 15 (17)
Oedema peripheral (General disorders) | 18 (19) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (5) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Weight increased (Investigations) | 4 (5) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 9 (9) | 6 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 0 (0)
Balance disorder (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 5 (5) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 9 (9) | 12 (12)
Headache (Nervous system disorders) | 3 (3) | 11 (11) | 7 (8)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 4 (5) | 2 (2)
Somnolence (Nervous system disorders) | 9 (9) | 8 (8) | 5 (5)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 17 (17) | 5 (5)
Sleep disorder (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (11) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 5 (5)
Hypertension (Vascular disorders) | 3 (3) | 7 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days